CLINICAL TRIAL: NCT00847132
Title: A Collaborative Care Program to Improve Depression Treatment in Cardiac Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jeff C. Huffman, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2007P-001152
Record Dates: First submitted 2009-02-17; First posted 2009-02-19 (Estimated); Results first posted 2017-03-31 (Actual); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Coronary Artery Disease; Congestive Heart Failure; Arrhythmia; Depression
Keywords: Collaborative Care
MeSH Terms: conditions — Coronary Artery Disease; Heart Failure; Arrhythmias, Cardiac; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Collaborative Care (Experimental): Collaborative Care Treatment: A study care manager provides depression education, consults with study psychiatrist to develop individualized treatment recommendations, and collaborates with patient and medical team to implement those recommendations
  Interventions: Behavioral: Collaborative Care Treatment
- Usual Care (Active Comparator): Usual Care Treatment: Primary medical providers are informed that the patient has depression and that treatment is recommended.
  Interventions: Behavioral: Usual Care Treatment

INTERVENTIONS:
Behavioral: Collaborative Care Treatment — Depression education, treatment recommendations, coordination of care
  Arms: Collaborative Care
Behavioral: Usual Care Treatment — Treatment as usual, providers are notified of diagnoses
  Arms: Usual Care

SUMMARY:
Depression in cardiac patients is common, persistent, and deadly. However, the vast majority of cardiac patients with depression go unrecognized and untreated, despite the existence of treatments that clearly improve depressive symptoms and may favorably impact survival. Our research group and others have found that depression recognition and treatment appears particularly limited among patients with acute cardiac illness, though this population may be the most vulnerable to the deleterious effects of depression. We propose a project, building on successful collaborative care depression management programs in outpatient settings, to address this important issue.

The specific hypotheses behind the proposed research are that a collaborative care depression management program can be successfully adapted to inpatient cardiac units, and that such a program will lead to greater rates of adequate depression treatment and improvements in secondary outcomes.

The following specific aims capture the stepwise goals of this program:

1. To determine whether a collaborative care depression management program ('Enhanced Care') leads to significantly increased rates of adequate depression treatment compared to usual care (screening and feedback) (Primary Aim).
2. To assess whether this Enhanced Care program has a lasting impact on adequate depression treatment, depressive symptoms, health-related quality of life, and adherence to medical recommendations at 6 weeks, 12 weeks, and 6 months, compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient admission for cardiac diagnosis
* Positive depression evaluation (PHQ-2>2, PHQ-9>9)
* Ability to provide informed consent

Exclusion Criteria:

* Active suicidal ideation
* Bipolar disorder, psychotic disorder, active substance use disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2007-07; Primary Completion 2010-01 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff C Huffman, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Sowden GL, Mastromauro CA, Seabrook RC, Celano CM, Rollman BL, Huffman JC. Baseline physical health-related quality of life and subsequent depression outcomes in cardiac patients. Psychiatry Res. 2013 Aug 15;208(3):288-90. doi: 10.1016/j.psychres.2013.05.019. Epub 2013 Jun 5. PMID 23747159
- [Derived] Bauer LK, Caro MA, Beach SR, Mastromauro CA, Lenihan E, Januzzi JL, Huffman JC. Effects of depression and anxiety improvement on adherence to medication and health behaviors in recently hospitalized cardiac patients. Am J Cardiol. 2012 May 1;109(9):1266-71. doi: 10.1016/j.amjcard.2011.12.017. Epub 2012 Feb 9. PMID 22325974
- [Derived] Celano CM, Mastromauro CA, Lenihan EC, Januzzi JL, Rollman BL, Huffman JC. Association of baseline anxiety with depression persistence at 6 months in patients with acute cardiac illness. Psychosom Med. 2012 Jan;74(1):93-9. doi: 10.1097/PSY.0b013e31823d38bc. Epub 2011 Dec 30. PMID 22210240
- [Derived] Huffman JC, Mastromauro CA, Sowden G, Fricchione GL, Healy BC, Januzzi JL. Impact of a depression care management program for hospitalized cardiac patients. Circ Cardiovasc Qual Outcomes. 2011 Mar;4(2):198-205. doi: 10.1161/CIRCOUTCOMES.110.959379. Epub 2011 Mar 8. PMID 21386067

RESULTS

PARTICIPANT FLOW:
Groups:
- Collaborative Care: A study care manager provides depression education, consults with study psychiatrist to develop individualized treatment recommendations, and collaborates with patient and medical team to implement those recommendations
  Collaborative care vs. usual care: depression education, treatment recommendations, coordination of care
- Usual Care: Primary medical providers are informed that the patient has depression and that treatment is recommended.
  Collaborative care vs. usual care: depression education, treatment recommendations, coordination of care
Period: Overall Study
Arm/Group | Collaborative Care | Usual Care
Started | 90 | 85
Completed | 89 | 84
Not Completed | 1 | 1
Not completed — Death | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Collaborative Care: A study care manager provides depression education, consults with study psychiatrist to develop individualized treatment recommendations, and collaborates with patient and medical team to implement those recommendations
  Collaborative Care Treatment: depression education, treatment recommendations, coordination of care
- Usual Care: Primary medical providers are informed that the patient has depression and that treatment is recommended.
  Usual Care Treatment: treatment as usual, providers are notified of diagnoses
- Total: Total of all reporting groups
Arm/Group | Collaborative Care | Usual Care | Total
Number analyzed (Participants) | 90 | 85 | 175
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (12.8) | 62.6 (12.2) | 62.35 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 47 | 85
  Male | 52 | 38 | 90
Race/Ethnicity, Customized [Number; unit: participants]
  White | 83 | 77 | 160
  Not White | 7 | 8 | 15
Region of Enrollment [Number; unit: participants]
  United States | 90 | 85 | 175
Patient Health Questionnaire-9 (PHQ-9) [Mean (Standard Deviation); unit: units on a scale] — The PHQ-9 is a 9-item scale that measures depression severity. Each question asks how often the subject experiences symptoms of depression and offers four answers: 0 = Not at all, 1 = Several days, 2 = More than half the days, 3 = Nearly every day. Scores are totaled and range from 0-27. To be considered depressed, subjects had to (a) have a total score of 10 or more, (b) answer five questions with a score of 2 or 3, and (c) one of the five questions had to be question 1 or question 2 (or both). Anyone who did not meet these criteria were not considered depressed.
  units on a scale | 17.9 (3.8) | 17.3 (3.1) | 17.6 (3.5)
Medical Outcomes Study Short Form-12 Mental Component Score (SF-12 MCS) [Mean (Standard Deviation); unit: units on a scale] — The SF-12 Mental Component Score is a 6-item scale that assesses mental health-related quality of life. Each question provides the option of 2-6 answers. Some questions are Yes/No (2 options), while others ask how often something occurs (6 options, etc.). Scores are calculated using a formula and can range from 0 to 100. A score of 50 indicates average mental health-related quality of life. Higher scores represent higher than average mental health-related quality of life, and lower scores represent lower mental health-related quality of life.
  units on a scale | 30.9 (8) | 32.5 (7.8) | 31.7 (7.9)
Hospital Anxiety and Depression Scale-Anxiety Subscale (HADS-A) [Mean (Standard Deviation); unit: units on a scale] — The HADS-A is a 7-item scale used to measure anxiety severity. Each question asks about a specific symptom of anxiety and offers four answers: 0 = Never / Not at all, 1 = A little / Time to time, 2 = Quite often / Usually, 3 = Most of the time / Very often. Scores are totaled and range from 0-21. A higher score means more anxiety.
  units on a scale | 10.8 (4.5) | 9.7 (4) | 10.3 (4.3)
Massachusetts General Hospital Cognitive and Physical Functioning Questionnaire (CPFQ) [Mean (Standard Deviation); unit: units on a scale] — The MGH CPFQ is a 7-item scale that assesses cognitive and executive function in mood and anxiety disorders. The MGH CPFQ asks about patients' abilities in different areas of cognition and executive function. Each question includes the following response options: 1 = greater than normal ability, 2 = normal ability, 3 = minimally diminished ability, 4 = moderately diminished ability, 5 = markedly diminished ability, 6 = totally absent ability. Scores are added and range from 7 to 42. Higher scores mean lower functioning abilities.
  units on a scale | 26.1 (5.2) | 25.4 (4.4) | 25.7 (4.8)
Women and Ischemia Syndrome Evaluation-Severity (WISE) [Mean (Standard Deviation); unit: units on a scale] — The WISE is a 10-item scale that assesses the number and severity of cardiac symptoms. Each question offers 4 responses: 0 = None (no symptom), 1 = Mild, 2 = Moderate, 3 = Severe.
  The "Severity" score represents the severity of cardiac illness. It's derived by adding all scores together. The Severity score can range from 0-30. A lower score means less severity of symptoms.
  The "Number" score represents the number of symptoms of cardiac illness. It's derived by counting the number of symptoms that scored 1 or more. The Number score can range from 0-10. A lower score means fewer symptoms.
  units on a scale | 12.1 (5.5) | 11.7 (4.6) | 11.9 (5.1)
Medical Outcomes Study Short Form-12 Physical Component Score (SF-12 PCS) [Mean (Standard Deviation); unit: units on a scale] — The SF-12 Physical Component Score is a 6-item scale that assesses physical health-related quality of life. Each question provides the option of 2-6 answers. Some questions are Yes/No (2 options), while others ask how often something occurs (6 options, etc.). Scores are calculated using a formula and can range from 0 to 100. A score of 50 indicates average physical health-related quality of life. Higher scores represent higher than average physical health-related quality of life, and lower scores represent lower physical health-related quality of life.
  units on a scale | 32.2 (10.4) | 31.3 (9.4) | 31.8 (9.9)
Women and Ischemia Syndrome Evaluation-Number (WISE) [Mean (Standard Deviation); unit: units on a scale] — The WISE is a 10-item scale that assesses the number and severity of cardiac symptoms. Each question offers 4 responses: 0 = None (no symptom), 1 = Mild, 2 = Moderate, 3 = Severe.
  The "Severity" score represents the severity of cardiac illness. It's derived by adding all scores together. The Severity score can range from 0-30. A lower score means less severity of symptoms.
  The "Number" score represents the number of symptoms of cardiac illness. It's derived by counting the number of symptoms that scored 1 or more. The Number score can range from 0-10. A lower score means fewer symptoms.
  units on a scale | 6.0 (2.2) | 6.1 (2.0) | 6.0 (2.1)

OUTCOME MEASURES:

1. Primary Outcome: Rates of Adequate Depression Treatment at Discharge
Description: Adequate treatment was defined a priori as either: (1) discharge prescription of an antidepressant at a clinically effective dose based on manufacturers' package labeling and treatment guidelines for the treatment of depression or (2) referral to a mental health treatment provider for psychotherapy (unless pre-planned as less than six sessions).
  Timeframe of "5 days after enrollment" was determined by calculating the median length of hospitalization for all subjects.
Time Frame: 5 days after enrollment
Measure: Number; unit: percentage of participants
Arm/Group | Collaborative Care | Usual Care
Number analyzed (Participants) | 89 | 84
percentage of participants | 71.9 | 9.5

2. Secondary Outcome: Change in Depression Symptoms From Baseline to 6 Months
Description: Depression symptoms measured by the Patient Health Questionnaire-9 (PHQ-9). The PHQ-9 is a 9-item scale that measures depression severity. Each question asks how often the subject experiences symptoms of depression and offers four answers: 0 = Not at all, 1 = Several days, 2 = More than half the days, 3 = Nearly every day. Scores are totaled and range from 0-27. To be considered depressed, subjects had to (a) have a total score of 10 or more, (b) answer five questions with a score of 2 or 3, and (c) one of the five questions had to be question 1 or question 2 (or both). Anyone who did not meet these criteria were not considered depressed.
Time Frame: Baseline, 6 weeks, 12 weeks, 6 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Collaborative Care | Usual Care
Number analyzed (Participants) | 89 | 84
units on a scale
  Baseline to 6 weeks | -8.98 [-10.26 to -7.70] | -5.95 [-7.40 to -4.50]
  6 weeks to 12 weeks | -8.73 [-10.06 to -7.38] | -5.30 [-6.75 to -3.85]
  12 weeks to 6 months | -8.67 [-10.17 to -7.16] | -6.90 [-8.20 to -5.59]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Collaborative Care | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/90 | 0/85
Other Adverse Events (participants affected / at risk) | 0/90 | 0/85

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No